CLINICAL TRIAL: NCT01933997
Title: A Phase 1 Study to Assess the Safety, Tolerability and Pharmacokinetics of Metadoxine (MG01CI) 1400 mg, Administered as Repeated Doses to Healthy Volunteers
Brief Title: A Phase 1 Study to Assess Pharmacokinetics of Metadoxine (MG01CI) 1400 mg, Administered to Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alcobra Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AL009
Record Dates: First submitted 2013-08-25; First posted 2013-09-04 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2013-10

CONDITIONS: Healthy Adult Subjects
Keywords: pharmacokinetics; metadoxine
MeSH Terms: interventions — metadoxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MG01CI 1400 mg (Experimental)
  Interventions: Drug: Metadoxine (MG01CI )

INTERVENTIONS:
Drug: Metadoxine (MG01CI )
  Other Names: MG01CI ,metadoxine

SUMMARY:
objective: To assess the safety, tolerability and pharmacokinetics of metadoxine, administered as repeated oral doses of MG01CI tablets (2 X 700 mg metadoxine per administration), to healthy adult subjects.

This is a single center, open-label, repeated-dose study in healthy male and female volunteers. Subjects will undergo screening within 21 days prior to the first dosing to assess their eligibility to participate in the study.

All subjects will receive 1400 mg metadoxine as two MG01CI oral extended-release tablets, administered once daily for five consecutive days.

Blood samples for metadoxine (which consists of two components: pyrrolidone-5-carboxylate and pyridoxine that can be identified in plasma concentration assays) will be drawn at designated time points, as described in the pharmacokinetic (PK) evaluation section. The subjects will remain confined to the unit for 6 days after first dosing.

A study termination visit will take place 10-12 days after the last dosing day. The subjects will be monitored for safety, and AEs (Adverse events) will be recorded throughout the study.

DETAILED DESCRIPTION:
This is a single center, open-label, repeated-dose study in healthy male and female volunteers. The overall study design is outlined in Figure 3.

Sixteen (16) healthy subjects will participate in the study (no less than 7 males and no less than 7 females).

The study will comprise a screening period (up to 21 days before first dosing), a dosing period in which the subjects will receive a daily single oral administration of 2 tablets, each containing 700 mg metadoxine (total of 1400 mg) for five consecutive days, and an EOS/Follow-up visit 10-12 days following the last dosing.

Subjects will be instructed to arrive at the CRC (clinical research center) clinic in the evening before the dosing period (Day 0). Check-in procedures will be performed as outlined in the Schedule of Events. The subjects will remain in the CRC for approximately 7 days.

Drugs will be administered after a 10-hour fast with 240 mL water. Drugs will be administered while the subjects are in bed sitting at an angle of at least 45 degrees, and, on Dosing Days 1 (first dosing) and 5 (last dosing) they will remain so for the next 4 hours.

There will be a 24-hour interval between each dosing. On Dosing Days 1 (first dosing) and 5 (last dosing) subjects will continue fasting for the next 4 hours post-dose, at which time a meal will be provided. Water will be allowed freely until one hour before, and from one hour after each dosing. Standardized meals will be provided according to the schedule Blood for PK analysis of metadoxine components (pyrrolidone-5-carboxylate L-pyroglutamic acid and pyridoxine) will be sampled serially following dosing as per the schedule in the PK Evaluation Subjects will be discharged from the CRC approximately 24 hours after the last dose.

There will be an end of study (EOS)/ follow-up visit to assess safety 10-12 days following the last dosing.

Analysis of the blood samples collected at the clinical facility to determine the plasma concentrations of metadoxine will be conducted by Avogadro, "Parc de Genibrat 31470 Fontenilles France".

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men and women between 18 and 45 years (inclusive) of age.
2. Subjects who provide written informed consent to participate in the study.
3. Body Mass Index (BMI) 19 to 29 kg/m2 (inclusive).
4. Non-smoking and no use of any tobacco or nicotine products (by declaration) for a period of at least 6 months prior to screening visit and a negative urine cotinine test which rules out active smoking at screening visit.
5. Subjects in general good health in the opinion of the investigator as determined by medical history, vital signs and a physical examination.
6. Blood pressure and heart rate within normal limits (blood pressure: systolic 90-140 mmHg; diastolic 50-90 mmHg, heart rate 50-100 beats per minute (bpm).
7. Female subjects must have a negative serum pregnancy test at screening and be willing and able to use a medically acceptable method of birth control or declare that they are abstaining from sexual intercourse, from the screening visit through the study termination visit or be surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) or post-menopausal. Postmenopausal women are defined as women with menstruation cessation for 12 consecutive months prior to signing of the informed consent form.
8. Electrocardiogram (ECG) with no clinically significant Investigator assessment discretion in cases of borderline results is allowed.
9. Negative HIV, Hepatitis B and Hepatitis C serology tests at screening.
10. No clinically significant abnormalities in hematology, blood chemistry, or urinalysis lab tests at screening.
11. No known history of alcohol or drug abuse. Negative urinary drugs of abuse screen determined within 21 days of the start of the study (Screening and check-in visit).
12. Subjects must be able to understand the requirements of the study and must be willing to comply with the requirements of the study.

Exclusion Criteria:

1. Known history of any significant medical disorder, which in the investigator's judgment contraindicates administration of the study medications.
2. Any clinically significant abnormality upon physical examination or in the clinical laboratory tests at screening visit.
3. Use of any prescription or over-the-counter (OTC) medications, including vitamins and herbal or dietary supplements within 14 days prior to first dosing. Paracetamol for symptomatic relief of pain is allowed until 24 hours prior to the first study drug administration.
4. Drug or alcohol abuse.
5. Known hypersensitivity and/or allergy to any drugs.
6. Any acute illness (e.g. acute infection) within 48 hours prior to the first study drug administration, which is considered of significance by the investigator.
7. Participation in another clinical trial with drugs received within 3 months prior to dosing (calculated from the previous study's last dosing date).
8. Subjects who donated blood in the three months or received blood or plasma derivatives in the six months preceding study drug administration.
9. Subjects with an inability to communicate well with the investigators and CRC staff (i.e., language problem, poor mental development or impaired cerebral function).
10. Inability to fast or consume the food provided in the study (including any known food allergies or food restrictions).
11. Pregnant or currently lactating women.
12. Subjects who are non-cooperative or unwilling to sign consent form

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2013-08; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) Endpoints | 6 weeks
  Pharmacokinetic calculations will be based on individual plasma concentrations of the blood sampling on Day 1 and Day 5.
  The following pharmacokinetic parameter will be calculated based on the plasma concentrations measured:
  Cmax Maximum concentration achieved
Pharmacokinetic (PK) Endpoints | 6 weeks
  The following pharmacokinetic parameter will be calculated based on the plasma concentrations measured:
  Tmax Time to reach maximum concentration (hours).
Pharmacokinetic (PK) Endpoints | 6 weeks
  The following pharmacokinetic parameter will be calculated based on the plasma concentrations measured:
  AUC (area under the curve) 0-t The area under the concentration vs. time curve, calculated as T1/2 Apparent terminal elimination half-life time (hours), The individual concentrations per time point will be displayed in graphs and listed per treatment day. Mean concentration per day and time point will be displayed graphically as well.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Atsmon, Dr., Principal Investigator — Souraski medical center
Locations (1):
- Clinical research center Souraski medical center, Tel Aviv, Israel